CLINICAL TRIAL: NCT05568511
Title: Home-based Digital Exercise Training Program to Improve Physical Function of Older Sepsis Survivors - HEAL Sepsis Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB202200027 -N-R; R21AG075645 (NIH); OCR42113 (Other: UF OnCore)
Record Dates: First submitted 2022-05-19; First posted 2022-10-05 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Exercise Program; Standard Care Control
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based, digitally delivered exercise training program (Experimental)
  Interventions: Other: App-based exercise program
- Standard care control group (Active Comparator)
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: App-based exercise program — Remotely-controlled, app-guided exercise program
  Arms: Home-based, digitally delivered exercise training program
Other: Standard of Care — These participants will follow the usual post-sepsis care after returning to home. The participants will be asked to log their daily activities in the app's health diary. The app will be activated for the baseline and follow-up physical function assessments, which will be supervised be a blinded coordinator via a video call.
  Arms: Standard care control group

SUMMARY:
Older sepsis survivors have poor physical function and need post-sepsis physical rehabilitation. Often times, sepsis survivors live far from research facilities and do not have access to rehabilitation services. Remotely delivered exercise intervention could be the key to improve physical function in this population. Therefore, the study proposes to recruit older sepsis survivors at discharge from the hospital to home and assign them to either exercise training or standard care.

DETAILED DESCRIPTION:
The proposed research will use a multi-disciplinary expertise of the University of Florida Sepsis and Critical Illness Research Center (SCIRC). For this project, the investigators will take advantage of the SCIRC's ongoing recruitment and monitoring of sepsis patients into an observational 1-year follow-up study. For this pilot, the investigators will approach and screen older sepsis survivors who get discharged from hospital to home. Potential participants will be approached within 5 days before discharge. The study will enroll 40 low-functioning (SPPB <6) older sepsis patients (≥55 years old). The enrolled subjects will be randomized to either digitally delivered and home-based exercise training program or standard care control group. All participants will receive tablets with the Blue Marble Health Platform (BMHP) app. For the control group, the app will be enabled only for the physical function assessments and for the rest of the time, only a health diary for logging daily activities will be available. Both groups will receive weekly phone calls from our research staff member to ask about their health and remind them of weekly charging of their tablets. The intervention group will receive daily reminders by text to perform the exercises for 30 min daily 5 days/week. Participants will be given wrist fitness tracking watches with step-counting and heart rate to measure adherence to an exercise intervention. At baseline and 12-week follow-up visits physical function assessments will be app-guided using the BMHP-validated physical function test similar to SPPB, with a blinded coordinator present via a video call to assist a participant with answering questions about the tests. The interventionists who will be calling the participants will be trained to maintain the same level of rapport to not jeopardize the study conditions.

ELIGIBILITY:
Inclusion Criteria:

* Able to perform lower and upper-body movements
* Sepsis survivor
* Age 55 years and older
* SPPB ≤ 6
* Being discharged to home from the hospital after surviving sepsis
* Willingness to be randomized to either treatment or control group
* Willingness to participate in all study procedures
* Willingness to use the devices and technology in the study

Exclusion Criteria:

* Failure to provide informed consent
* Pregnant
* Discharge to a long-term facility
* Involvement in a structured rehabilitation program
* Inability to perform lower or upper-body exercises (e.g. being in wheelchair)
* Severe cardiac disease, including NYHA Class III or IV congestive heart failure, clinically significant aortic stenosis, history of cardiac arrest, use of a cardiac defibrillator, or uncontrolled angina
* Significant cognitive impairment, including known dementia diagnosis or a Mini-Mental State Examination exam score < 24
* Progressive, degenerative neurologic disease, e.g., Parkinson's Disease, multiple sclerosis
* Severe pulmonary disease, requiring either steroid pills or injections or the use of supplemental oxygen
* Simultaneous participation in another intervention trial
* Poor or no cellular internet service at the primary place of living.

Ages: 55 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2025-07-29 (Actual); Study Completion 2025-07-29 (Actual)

PRIMARY OUTCOMES:
Feasibility (adherence - number of performed exercise sessions; retention - number of participants to complete the study). | Change from Baseline to 1 month and then 3 months
  Assessment of adherence (# of performed exercise sessions) and retention (# of participant that complete the study; # of completed days of the study).
Safety (number of adverse events) | Change from Baseline to 1 month and then 3 months
  Recording a number of adverse events during the study period.

SECONDARY OUTCOMES:
Physical function | Change from Baseline to 3 months
  Application-guided physical function testing. A test that assesses balance, walking speed and physical performance. Each item will be scored 0-4 (12 total). 0 being the worst and 12 being the best score. the Participants will perform it at their home with our blinded coordinator present via zoom.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Mankowski, PhD, Principal Investigator — University of Florida
Locations (1):
- UF Clinical and Translational Research Building, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zeidan RS, Ohama MK, Evripidou N, Anton SD, Hamed LL, Lin Y, Leeuwenburgh C, Guirguis FW, Efron PA, Flynn S, Smith B, Bacher R, Bakarasan N, Sarmiento Delgado J, Mankowski RT. Home-Based Digital Exercise Training Program to Improve Physical Function of Older Sepsis Survivors: Protocol of the HEAL Sepsis Randomized Clinical Trial. JMIR Res Protoc. 2024 Oct 17;13:e60270. doi: 10.2196/60270. PMID 39418096

DOCUMENTS (1):
  • Informed Consent Form (2025-01-07): https://cdn.clinicaltrials.gov/large-docs/11/NCT05568511/ICF_000.pdf